CLINICAL TRIAL: NCT02159976
Title: A Prospective, Multi-center, Randomized, Open-label, Parallel Design Clinical Trial to Compare 10-day Sequential Therapy and 14-day Modified Bismuth Quadruple Therapy for the Eradication of Helicobacter Pylori in Korea
Brief Title: Compare Sequential and Quadruple Therapy for the Eradication of Helicobacter Pylori in Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry); Chong Kun Dang Pharmaceutical (Industry); HK inno.N Corporation (Industry); Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, M.D, Ph.D., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1403/243-003
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Clarithromycin; Metronidazole; Tetracycline; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequential therapy (Active Comparator): pantoprazole 40mg bid 10 days (D1-D10), amoxicillin 1000mg bid 5 days (D1-D5), clarithromycin 500mg bid 5 days (D6-D10), metronidazole 500mg tid 5 days (D6-D10)
  Interventions: Drug: Pantoprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Metronidazole
- Modified bismuth quadruple therapy (Experimental): pantoprazole 40mg bid 14 days (D1-D14) , amoxicillin 1000mg bid 14 days (D1-D14), tetracycline 1000mg bid 14 days (D1-D14), bismuth 600mg bid 14 days (D1-D14)
  Interventions: Drug: Pantoprazole; Drug: Amoxicillin; Drug: Tetracycline; Drug: Bismuth

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole 40mg bid
Drug: Amoxicillin — Amoxicillin 1000mg bid
Drug: Clarithromycin — Clarithromycin 500mg bid
  Arms: Sequential therapy
Drug: Metronidazole — Metronidazole 500mg tid
  Arms: Sequential therapy
Drug: Tetracycline — Tetracycline 1000mg bid
  Arms: Modified bismuth quadruple therapy
Drug: Bismuth — Bismuth 600mg bid
  Arms: Modified bismuth quadruple therapy

SUMMARY:
1. To compare 10-day sequential therapy and 14-day modified bismuth quadruple therapy and to establish more effective first-line regimen for the eradication of Helicobacter pylori in Korea.
2. To evaluate the effect of H. pylori eradication therapy on the symptom improvement of functional dyspepsia

DETAILED DESCRIPTION:
Emerging evidence shows that the eradication rate of proton pump inhibitor (PPI)-based triple therapy for the first-line treatment of Helicobacter pylori has decreased. The reason for the decrease in the efficacy of PPI-based triple therapy is mainly due to the increase in the resistance against clarithromycin. Sequential therapy seems to be more effective than the PPI-based triple therapy, however, the eradication rate of sequential therapy in Korea, which is mostly under 80%, is still not satisfactory. Modified bismuth quadruple therapy which replace metronidazole with amoxicillin (contained PPI, bismuth, tetracycline and amoxicillin) can be a promising regimen because the antibiotic resistance rate of tetracycline and amoxicillin are relatively low in Korea and amoxicillin is more easy to take in comparing with metronidazole. Therefore, the aim of this study is to compare 10-day sequential therapy and 14-day modified bismuth quadruple therapy and to establish more effective first-line regimen for the eradication of Helicobacter pylori in Korea.

In addition, previous studies reported that H. pylori infection also associated with functional dyspepsia (FD) and recommended H. pylori eradication in patients with FD. However, until now, there was no randomized prospective study in Korea, therefore the another aim of this study is to evaluate the effect of H. pylori eradication therapy on the symptom improvement of FD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Korean Adult (Aged ≥ 18 years)
* Patients who diagnosis of H. pylori infection by any of following three methods

  * positive rapid urease test (CLOtest)
  * histologic evidence of H. pylori by modified Giemsa staining
  * positive 13C-urea breath test

Exclusion Criteria:

* Age under 18 years
* Previous eradication treatment for H. pylori
* Patients who took any drug which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics
* History of gastrectomy
* Advanced gastric cancer or other malignancy
* Abnormal liver function or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent diseases
* Previous allergic reactions to the study drugs
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee JY, Kim N, Park KS, Kim HJ, Park SM, Baik GH, Shim KN, Oh JH, Choi SC, Kim SE, Kim WH, Park SY, Kim GH, Lee BE, Jo Y, Hong SJ. Comparison of sequential therapy and amoxicillin/tetracycline containing bismuth quadruple therapy for the first-line eradication of Helicobacter pylori: a prospective, multi-center, randomized clinical trial. BMC Gastroenterol. 2016 Jul 26;16(1):79. doi: 10.1186/s12876-016-0490-8. PMID 27460100

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Therapy: pantoprazole 40mg bid 10 days (D1-D10), amoxicillin 1000mg bid 5 days (D1-D5), clarithromycin 500mg bid 5 days (D6-D10), metronidazole 500mg tid 5 days (D6-D10)
  Pantoprazole
  Amoxicillin
  Clarithromycin
  Metronidazole
- Modified Bismuth Quadruple Therapy: pantoprazole 40mg bid 14 days (D1-D14) , amoxicillin 1000mg bid 14 days (D1-D14), tetracycline 1000mg bid 14 days (D1-D14), bismuth 600mg bid 14 days (D1-D14)
  Pantoprazole
  Amoxicillin
  Tetracycline
  Bismuth
Period: Overall Study
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy
Started | 195 | 195
Completed | 165 | 170
Not Completed | 30 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy | Total
Number analyzed (Participants) | 195 | 195 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 154 | 150 | 304
  >=65 years | 41 | 45 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.6) | 53.6 (13.2) | 53.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 78 | 170
  Male | 103 | 117 | 220
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 195 | 195 | 390

OUTCOME MEASURES:

1. Primary Outcome: Counts of Participants With Successful H. Pylori Eradication
Time Frame: 4 weeks after termination of eradication therapy, up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy
Number analyzed (Participants) | 195 | 195
Participants | 146 | 134

2. Secondary Outcome: Counts of Participants Whose Drug Compliance is More Than 85%
Time Frame: 4 weeks after termination of eradication therapy, up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy
Number analyzed (Participants) | 176 | 177
Participants | 165 | 170

3. Secondary Outcome: Counts of Participants With Adverse Event
Time Frame: 4 weeks after termination of eradication therapy, up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy
Number analyzed (Participants) | 195 | 195
Participants | 93 | 72

4. Secondary Outcome: Functional Dyspepsia Symptom Responses Rate
Time Frame: 1 year after termination of eradication therapy
Population: SQT and PBAT were used for the initial treatment. Thereafter, treatment success and treatment failure group were divided. In the treatment failure group, secondary treatment was performed. Secondary endpoints were functional and dyspepsia symptom responses rate after successful treatment, not success in both treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- In Eradication Success Group: functional dyspepsia symptom responses rate in eradication success group
- In Eradication Failure Group: functional dyspepsia symptom responses rate in eradication failure group
Arm/Group | In Eradication Success Group | In Eradication Failure Group
Number analyzed (Participants) | 60 | 3
Participants
  complete (≥75%) | 44 | 0
  Satisfactory (50-74%) | 1 | 0
  Partial (25-49%) | 6 | 1
  Refractory (<25%) | 9 | 2

ADVERSE EVENTS:
Arm/Group | Sequential Therapy | Modified Bismuth Quadruple Therapy
Serious Adverse Events (participants affected / at risk) | 0/195 | 0/195
Other Adverse Events (participants affected / at risk) | 93/195 | 72/195
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sequential Therapy (N=195) | Modified Bismuth Quadruple Therapy (N=195)
Bloating (Gastrointestinal disorders) | 21 | 11
Epigastric soreness (Gastrointestinal disorders) | 15 | 17
Taste distortions (Gastrointestinal disorders) | 24 | 4
Nausea (Gastrointestinal disorders) | 14 | 6
Anorexia (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Headache (Nervous system disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 12
Constipation (Gastrointestinal disorders) | 2 | 3
Reflux (Gastrointestinal disorders) | 1 | 1
Rash and itching (Skin and subcutaneous tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 1 | 0
Stool color change (Gastrointestinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No